CLINICAL TRIAL: NCT05014282
Title: Randomized Trial of Automated Video-Assisted Smoking Treatment for People Living With HIV (Project RESOURCE)
Brief Title: Automated Video-Assisted Smoking Treatment for People Living With HIV
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MCC-20262; R01CA243552 (NIH)
Record Dates: First submitted 2021-08-13; First posted 2021-08-20 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Tobacco Use Cessation Devices; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Treatment (Active Comparator): Participants randomized to Standard Treatment (ST) will be provided with a 10-week supply of nicotine patches and lozenges. ST participants will be connected with their state's tobacco quitline services and will complete weekly 4-item smartphone assessments electronically for 26 weeks. The weekly assessments consist of questions on smoking status, motivation, self-efficacy, and perceived stress.
  Interventions: Drug: Nicotine patch; Behavioral: Counseling; Drug: Nicotine lozenge
- Automated Treatment (Experimental): Participants randomized to Automated Treatment (AT) will be given a 10-week supply of nicotine patches and lozenges. AT will also comprise of: 1) 12 proactive treatment videos, delivered weekly, that are tailored on smoking status, motivation, agency, and/or negative affect/stress; 2) 26 weeks of on-demand access to treatment content; 3) 26 weeks of text content
  Interventions: Drug: Nicotine patch; Drug: Nicotine lozenge; Behavioral: Smartphone-delivered automated treatment

INTERVENTIONS:
Drug: Nicotine patch — Participants will be provided with a 10-week supply of nicotine patches
Behavioral: Counseling — Phone counseling with the state tobacco quitline.
  Arms: Standard Treatment
Drug: Nicotine lozenge — Participants will be provided with a 10-week supply of nicotine lozenges
Behavioral: Smartphone-delivered automated treatment — An interactive smartphone-based intervention that comprises content delivered via audio/video clips and text content automatically each week to the participant
  Arms: Automated Treatment

SUMMARY:
This study will evaluate if Automated Treatment performs better, in terms of facilitating long-term smoking abstinence, than the more resource-intensive Standard Treatment.

ELIGIBILITY:
Inclusion Criteria:

* smoked >/=100 cigarettes in lifetime
* English or Spanish speaking
* Currently smoke > 5 cigarettes/day
* Willing to make a quit attempt within 1 week of enrollment
* HIV positive
* Process a smartphone compatible with the project app
* Have a valid email address

Exclusion Criteria:

* Currently pregnant or breastfeeding
* Current use of smoking cessation medications
* Enrolled in a smoking cessation study
* Household member enrolled in the study
* Failure to electronically confirm participation within 14 days of randomization via electronic link sent to participant's smartphone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 638 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2025-09-23 (Actual); Study Completion 2026-09-23 (Estimated)

PRIMARY OUTCOMES:
Self Reported 7 Day Abstinence Smoking Status | 12 Month Follow-Up
  Participants will self report 7-day abstinence smoking status

SECONDARY OUTCOMES:
Smoking Status by Saliva Cotinine Kit | 12 Month Follow-Up
  Investigators will verify smoking status by collecting cotinine sample from a saliva cotinine kit.
Self Reported 24 Hours Smoking Abstinence | 12 Month Follow-Up
  Number of participants who report they quit smoking for 24 hours
30 Day Smoking Abstinence | 12 Month Follow-Up
  Number of participants who report they quit smoking for 30 days
Continuous Smoking Abstinence | 12 Month Follow-Up
  Number of participants who report they quit smoking

CONTACTS AND LOCATIONS:
Overall Officials: Damon J Vidrine, Dr.PH, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vidrine DJ, Bui TC, Businelle MS, Shih YT, Sutton SK, Shahani L, Hoover DS, Bowles K, Vidrine JI. Evaluating the Efficacy of Automated Smoking Treatment for People With HIV: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2021 Nov 17;10(11):e33183. doi: 10.2196/33183. PMID 34787590
- See also: Moffitt Clinical Trial Search — https://moffitt.org/clinical-trials-research/clinical-trials/